CLINICAL TRIAL: NCT04311619
Title: Does Repetitive Transcranial Magnetic Stimulation (rTMS) Induce Synaptic Plasticity?
Brief Title: Does rTMS Induce Synaptic Plasticity?
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: We did not receive grant funding for this study.
Sponsor: Davidzon, Guido, M.D. (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Jong Yoon, Associate Professor of Psychiatry and Behavioral Sciences, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 54574
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Major Depression Disorder Participants (Experimental): Participants will undergo positron emission tomography-magnetic resonance (PET-MR) imaging using the [11C]UCB-J radiotracer before and after Repetitive Transcranial Magnetic Stimulation (rTMS) treatment
  Interventions: Drug: [11C]UCB-J radiotracer; Device: PET-MR

INTERVENTIONS:
Drug: [11C]UCB-J radiotracer — I.V. bolus administration of up to 15 mCi (equivalent to 0.3 rems) in the antecubital vein per injection
  Other Names: C11-UCB-J
Device: PET-MR — Positron emission tomography and magnetic resonance imaging, with a scan duration of up to 120 minutes

SUMMARY:
The purpose of this study is to utilize the radioactive positron emission tomography (PET) tracer [11C]UCB-J to investigate the effect of repetitive transcranial magnetic stimulation (rTMS) on synaptic plasticity. UCB-J has been validated as a marker for synaptic density. We will use this tracer to examine if rTMS leads to changes in synaptic plasticity, specifically changes in synaptic density, in individuals receiving rTMS for MDD. If rTMS is proven effective for increasing synaptic plasticity, there is a significant potential of a new applicable treatment for a variety of diseases that affect brain physiology.

DETAILED DESCRIPTION:
The objective of this project is to discover the neural mechanisms by which Major Depressive Disorder (MDD) is treated, so that we may gain insights into its pathophysiology, as well as to develop new biomarkers. We will utilize the PET tracer [11C]UCB-J, the first in human tracer of neural synapses, to test the hypothesis that the successful treatment of MDD with repetitive Transcranial Magnetic Stimulation (rTMS) is associated with increased synaptic density. We will use this tracer to measure synaptic density before and after rTMS treatment and compare change in synaptic density between subjects who respond to the rTMS treatment and those who do not respond to treatment.

The finding of a marked increase in synaptic density in participants who respond to rTMS treatment would point to the possibility of developing new treatments with the potential to modify disease through mitigating, preventing or remediating synaptic loss.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years in age
* U.S. Veteran
* Diagnosis of MDD
* On a stable medication regimen for at least two weeks prior to testing
* Stable social environment and housing to enable regular attendance at clinic visits
* Ability to undergo cognitive testing, clinical assessments, and PET/MR scans
* Stable medical health
* Will undergo rTMS treatment for MDD at the VA Palo Alto
* Able to complete a PET-MR scan without the use of sedation

Exclusion Criteria:

* Active substance use within three months of testing
* IQ < 70
* Major medical neurological illness or significant head trauma
* Pregnancy or breastfeeding
* Contraindication to MR scanning, including magnetic-resonance incompatible metal or hardware including pacemakers, cochlear implants, and bullets near a critical organ
* Weight > 350 lbs or a large body habitus that MR scanner cannot accommodate
* History of or current claustrophobia
* Inability to comply with basic study requirements such as following directions and punctuality
* Acute or unstable chronic medical illness that would affect participation or compliance with study procedures, e.g. unstable angina
* Unstable psychiatric symptoms that precludes consistent participation in the study, e.g. active current suicidal intent or plan, severe psychosis
* Inability to undergo PET/MR scan, e.g. claustrophobia, presence of ferromagnetic objects in subject's body

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Synaptic Density Quantified by Regional Binding Potential (BP_ND) | Assessed during PET scans before and after rTMS therapy (90 minutes per scan)
  Synaptic density change (Baseline minus Post Treatment) will be quantified between treatment responsive patients and treatment unresponsive patients with the regional binding potential (BP_ND), a measure of [11C]UCB-J binding. BP_ND will be derived by using the simplified reference tissue model and the centrum semiovale as the reference region. This method has been recently utilized by other investigators in neuropsychiatric samples. Both exploratory voxel-wise BP_ND and region of interest (ROI) BP_ND will be compared across groups. ROIs include the striatum, dorsolateral prefrontal cortex, hippocampus, and superior temporal cortex.

CONTACTS AND LOCATIONS:
Overall Officials: Jong H Yoon, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - VA Palo Alto Health Care System, Palo Alto, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No
No current plan to share data

REFERENCES:
- [Background] Finnema SJ, Nabulsi NB, Mercier J, Lin SF, Chen MK, Matuskey D, Gallezot JD, Henry S, Hannestad J, Huang Y, Carson RE. Kinetic evaluation and test-retest reproducibility of [11C]UCB-J, a novel radioligand for positron emission tomography imaging of synaptic vesicle glycoprotein 2A in humans. J Cereb Blood Flow Metab. 2018 Nov;38(11):2041-2052. doi: 10.1177/0271678X17724947. Epub 2017 Aug 9. PMID 28792356
- [Background] Chen MK, Mecca AP, Naganawa M, Finnema SJ, Toyonaga T, Lin SF, Najafzadeh S, Ropchan J, Lu Y, McDonald JW, Michalak HR, Nabulsi NB, Arnsten AFT, Huang Y, Carson RE, van Dyck CH. Assessing Synaptic Density in Alzheimer Disease With Synaptic Vesicle Glycoprotein 2A Positron Emission Tomographic Imaging. JAMA Neurol. 2018 Oct 1;75(10):1215-1224. doi: 10.1001/jamaneurol.2018.1836. PMID 30014145
- [Background] Wu Y, Carson RE. Noise reduction in the simplified reference tissue model for neuroreceptor functional imaging. J Cereb Blood Flow Metab. 2002 Dec;22(12):1440-52. doi: 10.1097/01.WCB.0000033967.83623.34. PMID 12468889
- [Background] Chervyakov AV, Chernyavsky AY, Sinitsyn DO, Piradov MA. Possible Mechanisms Underlying the Therapeutic Effects of Transcranial Magnetic Stimulation. Front Hum Neurosci. 2015 Jun 16;9:303. doi: 10.3389/fnhum.2015.00303. eCollection 2015. PMID 26136672
- [Background] Holmes SE, Scheinost D, Finnema SJ, Naganawa M, Davis MT, DellaGioia N, Nabulsi N, Matuskey D, Angarita GA, Pietrzak RH, Duman RS, Sanacora G, Krystal JH, Carson RE, Esterlis I. Lower synaptic density is associated with depression severity and network alterations. Nat Commun. 2019 Apr 4;10(1):1529. doi: 10.1038/s41467-019-09562-7. PMID 30948709